CLINICAL TRIAL: NCT01876823
Title: Effects of Combined Memantine (Namenda) Plus Escitalopram (Lexapro) Treatment in Elderly Depressed Patients With Cognitive Impairment
Brief Title: Memantine Plus Es-citalopram in Elderly Depressed Patients With Cognitive Impairment
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6277R
Record Dates: First submitted 2013-06-05; First posted 2013-06-13 (Estimated); Results first posted 2014-10-24 (Estimated); Last update posted 2014-10-24 (Estimated); Status verified 2013-09

CONDITIONS: Mild Cognitive Impairment; Major Depressive Disorder; Alzheimer's Disease
Keywords: Memory Decline; Depression; Elderly; Antidepressants; Treatment; memantine
MeSH Terms: conditions — Cognitive Dysfunction; Depressive Disorder, Major; Alzheimer Disease; Depression | interventions — Escitalopram; Memantine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- es-citalopram and Memantine Treatment (Experimental): concurrent es-citalopram plus memantine were administered for 48 weeks.
  Interventions: Drug: es-citalopram; Drug: Memantine

INTERVENTIONS:
Drug: es-citalopram — es-citalopram 10mg/day will be given for the first week, and 20mg/day starting at week 2.
  Other Names: Lexapro
Drug: Memantine — After two weeks on Lexapro, Memantine 5mg will be added. The dose will increase to 10mg for the second week and will be increased at a rate of 5mg per week. Memantine dosage will not exceed 20mg.
  Other Names: Namenda

SUMMARY:
Alzheimer's disease (AD), the most common dementing disorder of later life, is a major cause of disability and death in the elderly. Although a number of theoretical causes exist, the etiology of AD is still unknown. Consequently, the focus of treatments has been palliative, designed to ameliorate AD symptoms. Recent efforts, however, have revealed some surprising data suggesting that cholinesterase inhibitors (AchEIs), used over the last decade, and recently released memantine (an N-methyl-D-aspartate (NMDA) receptor antagonist), may confer protection to neurons. Thus, they may offer a slowing of cognitive decline and/or improvement in behavioral symptoms associated with memory impairment.

Over the last decade, it has been well documented that mild cognitive impairment (MCI) increases the risk of conversion to AD and that coincident depression and MCI (Dep-MCI) further increases the risk 2 to 3 fold. The primary focus of this line of investigation is to treat the very high risk to dement patient population with Dep-MCI, before they develop AD, in the hopes of delaying AD onset.

Memantine had not been studied in DEP-MCI patients. Since treatment of these patients with combined antidepressant and AChEIs has been associated with cognitive improvement in pilot studies, we explore whether treatment of DEP-MCI with memantine in addition to antidepressant treatment would benefit cognitive performance and lead to a low rate of conversion to dementia. We evaluate the cognitive and antidepressant benefit of combined open-label es-citalopram and memantine treatment over 48 weeks in a DEP-CI sample.

DETAILED DESCRIPTION:
The study is conducted in a sample of 35 elderly (50-90 years old) outpatients who meet study inclusion criteria for depression (DEP) (DSM-IV criteria for major depression, dysthymic disorder, or depression NOS) and mild cognitive impairment (MCI; e.g. operationally defined as between "normal" and "dementia"), i.e., Dep-MCI. The research plan includes: i) Obtaining a baseline psychiatric and neuropsychological test profile, ii) If currently on an ineffective antidepressant, having a one week washout (3 weeks for fluoxetine), iii) A treatment trial beginning with a two-week es-citalopram lead-in period. At two weeks, memantine (Namenda) is added starting at 5 mg/day and increased until the maximum dose of 20 mg/day is reached by six weeks. The study psychiatrist administers: the 24-item Hamilton Depression Rating Scale (HAM-D); the Clinical Global Impression (CGI, 1-7 scale) initial severity and subsequent change ratings separately for depression, cognition, and overall clinical status; the Treatment Emergent Symptom Scale (TESS) for somatic side effects. A trained technician administers the neuropsychological battery at baseline, 12, 24 and 48 weeks. If the patient is an antidepressant non-responder during the first 12-weeks, the es-citalopram is changed to an alternative antidepressant, as clinically indicated by the treating psychiatrist. The patient remains on the memantine for the entire 48-weeks, irrespective of antidepressant response.

This will tell us about the efficacy and tolerability of es-citalopram+memantine on both cognitive and depressive symptoms in Dep-MCI patients and will potentially have broader public health implications because Dep-MCI is a wide-spread clinical problem where management needs to be improved.

ELIGIBILITY:
Inclusion Criteria:

1. Of either sex, age greater than 49 years old
2. Meets criteria for both "depression" and "cognitive impairment".
3. Study Criteria for "depression":

   i. Patients who meet DSM-IV criteria for Major Depression, Dysthymic Disorder, or Dysthymia symptoms criteria of minimum 6 month duration (not the 2 year DSM-IV criteria). ii. 24-item HAM-D greater than 13; and iii. Clinical Global Impression (CGI) for severity of Depression greater than 2 (absolute score at least mild to moderate depression on a 7-point scale)
4. Study Criteria for "cognitive deficit":

   i. Subjective memory complaint ii.Mini Mental Status Exam (MMSE) greater than 24; and at least one of a, b, or c:
   1. less than 3 on MMSE 5 min delay on recall
   2. scores on 2 neuropsychological tests greater than 1 Standard Deviation (SD) below standardized norms, or
   3. score on 1 neuropsychological tests greater than 2 SD below standardized norms.

   Neuropsychological tests for inclusion criteria (subset of larger battery):

   Selective Reminding Test with delay Wechsler Memory Scale (WMS): Visual Reproduction - with delay, % savings from immed to delay Controlled Oral Word Association Test Trails B Digit symbol subtest of Wechsler Adult Intelligence Scale (WAIS)-III Continuous Performance Test iii. CGI for severity of Cognitive deficit greater than 2 (absolute score on a 7-point scale:1=no deficit to 7=severe deficit). iv. Clinical Dementia Rating (CDR) = 0 or 0.5
5. Willing and capable of giving informed consent

Exclusion Criteria:

1. Meets Criteria for dementia (DSM-IV) or probable Alzheimer's disease by National Institute of Neurological and Communicative Disorders and Stroke and the Alzheimer's Disease and Related Disorders Association criteria (NINCDS-ADRDA criteria)
2. Meets criteria for:

   1. schizophrenia
   2. alcohol or substance dependence or abuse within the last 6 months.
3. Suicidal attempt in last 6 months or current suicidal intent.
4. Patients currently on an effective antidepressant medication
5. Use of cholinesterase inhibitors in the last year.
6. Neurological disease including stroke, epilepsy, or other neurodegenerative disorders.
7. An acute, severe or unstable medical condition such as metastatic or active cancer, hepatic disease, or primary renal disease requiring dialysis.
8. Patients who can not tolerate being tapered off antidepressant medication (i.e. greater than a 25% incr. in baseline HAM-D) or has a history indicating patient is unlikely to tolerate psychotropic washout.
9. Patient with a history of non-response to Citalopram or es-citalopram

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2006-04; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Pelton, M.D., Principal Investigator — New York State Psychiatric Institute; Davangere Devanand, M.D., Study Chair — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

REFERENCES:
- [Background] Alexopoulos GS, Meyers BS, Young RC, Mattis S, Kakuma T. The course of geriatric depression with "reversible dementia": a controlled study. Am J Psychiatry. 1993 Nov;150(11):1693-9. doi: 10.1176/ajp.150.11.1693. PMID 8105707
- [Background] Atri A, Shaughnessy LW, Locascio JJ, Growdon JH. Long-term course and effectiveness of combination therapy in Alzheimer disease. Alzheimer Dis Assoc Disord. 2008 Jul-Sep;22(3):209-21. doi: 10.1097/WAD.0b013e31816653bc. PMID 18580597
- [Background] Bakchine S, Loft H. Memantine treatment in patients with mild to moderate Alzheimer's disease: results of a randomised, double-blind, placebo-controlled 6-month study. J Alzheimers Dis. 2008 Feb;13(1):97-107. doi: 10.3233/jad-2008-13110. PMID 18334761
- [Background] Barnes DE, Yaffe K, Byers AL, McCormick M, Schaefer C, Whitmer RA. Midlife vs late-life depressive symptoms and risk of dementia: differential effects for Alzheimer disease and vascular dementia. Arch Gen Psychiatry. 2012 May;69(5):493-8. doi: 10.1001/archgenpsychiatry.2011.1481. PMID 22566581
- [Background] Bassuk SS, Berkman LF, Wypij D. Depressive symptomatology and incident cognitive decline in an elderly community sample. Arch Gen Psychiatry. 1998 Dec;55(12):1073-81. doi: 10.1001/archpsyc.55.12.1073. PMID 9862549
- [Background] Boyle PA, Wilson RS, Aggarwal NT, Tang Y, Bennett DA. Mild cognitive impairment: risk of Alzheimer disease and rate of cognitive decline. Neurology. 2006 Aug 8;67(3):441-5. doi: 10.1212/01.wnl.0000228244.10416.20. PMID 16894105
- [Background] Burt DB, Zembar MJ, Niederehe G. Depression and memory impairment: a meta-analysis of the association, its pattern, and specificity. Psychol Bull. 1995 Mar;117(2):285-305. doi: 10.1037/0033-2909.117.2.285. PMID 7724692
- [Background] Charney DS, Reynolds CF 3rd, Lewis L, Lebowitz BD, Sunderland T, Alexopoulos GS, Blazer DG, Katz IR, Meyers BS, Arean PA, Borson S, Brown C, Bruce ML, Callahan CM, Charlson ME, Conwell Y, Cuthbert BN, Devanand DP, Gibson MJ, Gottlieb GL, Krishnan KR, Laden SK, Lyketsos CG, Mulsant BH, Niederehe G, Olin JT, Oslin DW, Pearson J, Persky T, Pollock BG, Raetzman S, Reynolds M, Salzman C, Schulz R, Schwenk TL, Scolnick E, Unutzer J, Weissman MM, Young RC; Depression and Bipolar Support Alliance. Depression and Bipolar Support Alliance consensus statement on the unmet needs in diagnosis and treatment of mood disorders in late life. Arch Gen Psychiatry. 2003 Jul;60(7):664-72. doi: 10.1001/archpsyc.60.7.664. PMID 12860770
- [Background] Chen X, Magnotta VA, Duff K, Boles Ponto LL, Schultz SK. Donepezil effects on cerebral blood flow in older adults with mild cognitive deficits. J Neuropsychiatry Clin Neurosci. 2006 Spring;18(2):178-85. doi: 10.1176/jnp.2006.18.2.178. PMID 16720794
- [Background] Culang ME, Sneed JR, Keilp JG, Rutherford BR, Pelton GH, Devanand DP, Roose SP. Change in cognitive functioning following acute antidepressant treatment in late-life depression. Am J Geriatr Psychiatry. 2009 Oct;17(10):881-8. doi: 10.1097/jgp.0b013e3181b4bf4a. PMID 19916207
- [Background] Devanand DP, Liu X, Tabert MH, Pradhaban G, Cuasay K, Bell K, de Leon MJ, Doty RL, Stern Y, Pelton GH. Combining early markers strongly predicts conversion from mild cognitive impairment to Alzheimer's disease. Biol Psychiatry. 2008 Nov 15;64(10):871-9. doi: 10.1016/j.biopsych.2008.06.020. Epub 2008 Aug 23. PMID 18723162
- [Background] Devanand DP, Pelton GH, Marston K, Camacho Y, Roose SP, Stern Y, Sackeim HA. Sertraline treatment of elderly patients with depression and cognitive impairment. Int J Geriatr Psychiatry. 2003 Feb;18(2):123-30. doi: 10.1002/gps.802. PMID 12571820
- [Background] Devanand DP, Sano M, Tang MX, Taylor S, Gurland BJ, Wilder D, Stern Y, Mayeux R. Depressed mood and the incidence of Alzheimer's disease in the elderly living in the community. Arch Gen Psychiatry. 1996 Feb;53(2):175-82. doi: 10.1001/archpsyc.1996.01830020093011. PMID 8629893
- [Background] Doody RS, Ferris SH, Salloway S, Sun Y, Goldman R, Watkins WE, Xu Y, Murthy AK. Donepezil treatment of patients with MCI: a 48-week randomized, placebo-controlled trial. Neurology. 2009 May 5;72(18):1555-61. doi: 10.1212/01.wnl.0000344650.95823.03. Epub 2009 Jan 28. PMID 19176895
- [Background] Farrimond LE, Roberts E, McShane R. Memantine and cholinesterase inhibitor combination therapy for Alzheimer's disease: a systematic review. BMJ Open. 2012 Jun 11;2(3):e000917. doi: 10.1136/bmjopen-2012-000917. Print 2012. PMID 22689908
- [Background] Feldman HH, Ferris S, Winblad B, Sfikas N, Mancione L, He Y, Tekin S, Burns A, Cummings J, del Ser T, Inzitari D, Orgogozo JM, Sauer H, Scheltens P, Scarpini E, Herrmann N, Farlow M, Potkin S, Charles HC, Fox NC, Lane R. Effect of rivastigmine on delay to diagnosis of Alzheimer's disease from mild cognitive impairment: the InDDEx study. Lancet Neurol. 2007 Jun;6(6):501-12. doi: 10.1016/S1474-4422(07)70109-6. PMID 17509485
- [Background] Ferris S, Schneider L, Farmer M, Kay G, Crook T. A double-blind, placebo-controlled trial of memantine in age-associated memory impairment (memantine in AAMI). Int J Geriatr Psychiatry. 2007 May;22(5):448-55. doi: 10.1002/gps.1711. PMID 17117395
- [Background] Fischer P, Jungwirth S, Zehetmayer S, Weissgram S, Hoenigschnabl S, Gelpi E, Krampla W, Tragl KH. Conversion from subtypes of mild cognitive impairment to Alzheimer dementia. Neurology. 2007 Jan 23;68(4):288-91. doi: 10.1212/01.wnl.0000252358.03285.9d. PMID 17242334
- [Background] Gabryelewicz T, Styczynska M, Luczywek E, Barczak A, Pfeffer A, Androsiuk W, Chodakowska-Zebrowska M, Wasiak B, Peplonska B, Barcikowska M. The rate of conversion of mild cognitive impairment to dementia: predictive role of depression. Int J Geriatr Psychiatry. 2007 Jun;22(6):563-7. doi: 10.1002/gps.1716. PMID 17136705
- [Background] Green RC, Cupples LA, Kurz A, Auerbach S, Go R, Sadovnick D, Duara R, Kukull WA, Chui H, Edeki T, Griffith PA, Friedland RP, Bachman D, Farrer L. Depression as a risk factor for Alzheimer disease: the MIRAGE Study. Arch Neurol. 2003 May;60(5):753-9. doi: 10.1001/archneur.60.5.753. PMID 12756140
- [Background] Grober E, Lipton RB, Hall C, Crystal H. Memory impairment on free and cued selective reminding predicts dementia. Neurology. 2000 Feb 22;54(4):827-32. doi: 10.1212/wnl.54.4.827. PMID 10690971
- [Background] Houde M, Bergman H, Whitehead V, Chertkow H. A predictive depression pattern in mild cognitive impairment. Int J Geriatr Psychiatry. 2008 Oct;23(10):1028-33. doi: 10.1002/gps.2028. PMID 18651723
- [Background] Koontz J, Baskys A. Effects of galantamine on working memory and global functioning in patients with mild cognitive impairment: a double-blind placebo-controlled study. Am J Alzheimers Dis Other Demen. 2005 Sep-Oct;20(5):295-302. doi: 10.1177/153331750502000502. PMID 16273995
- [Background] Lange KL, Bondi MW, Salmon DP, Galasko D, Delis DC, Thomas RG, Thal LJ. Decline in verbal memory during preclinical Alzheimer's disease: examination of the effect of APOE genotype. J Int Neuropsychol Soc. 2002 Nov;8(7):943-55. doi: 10.1017/s1355617702870096. PMID 12405546
- [Background] Lopez OL, Becker JT, Wahed AS, Saxton J, Sweet RA, Wolk DA, Klunk W, Dekosky ST. Long-term effects of the concomitant use of memantine with cholinesterase inhibition in Alzheimer disease. J Neurol Neurosurg Psychiatry. 2009 Jun;80(6):600-7. doi: 10.1136/jnnp.2008.158964. Epub 2009 Feb 9. PMID 19204022
- [Background] Lu PH, Edland SD, Teng E, Tingus K, Petersen RC, Cummings JL; Alzheimer's Disease Cooperative Study Group. Donepezil delays progression to AD in MCI subjects with depressive symptoms. Neurology. 2009 Jun 16;72(24):2115-21. doi: 10.1212/WNL.0b013e3181aa52d3. PMID 19528519
- [Background] Manly JJ, Tang MX, Schupf N, Stern Y, Vonsattel JP, Mayeux R. Frequency and course of mild cognitive impairment in a multiethnic community. Ann Neurol. 2008 Apr;63(4):494-506. doi: 10.1002/ana.21326. PMID 18300306
- [Background] McShane R, Areosa Sastre A, Minakaran N. Memantine for dementia. Cochrane Database Syst Rev. 2006 Apr 19;(2):CD003154. doi: 10.1002/14651858.CD003154.pub5. PMID 16625572
- [Background] Modrego PJ, Ferrandez J. Depression in patients with mild cognitive impairment increases the risk of developing dementia of Alzheimer type: a prospective cohort study. Arch Neurol. 2004 Aug;61(8):1290-3. doi: 10.1001/archneur.61.8.1290. PMID 15313849
- [Background] Morris JC, Storandt M, Miller JP, McKeel DW, Price JL, Rubin EH, Berg L. Mild cognitive impairment represents early-stage Alzheimer disease. Arch Neurol. 2001 Mar;58(3):397-405. doi: 10.1001/archneur.58.3.397. PMID 11255443
- [Background] Nyakas C, Granic I, Halmy LG, Banerjee P, Luiten PG. The basal forebrain cholinergic system in aging and dementia. Rescuing cholinergic neurons from neurotoxic amyloid-beta42 with memantine. Behav Brain Res. 2011 Aug 10;221(2):594-603. doi: 10.1016/j.bbr.2010.05.033. Epub 2010 May 27. PMID 20553766
- [Background] Ownby RL, Crocco E, Acevedo A, John V, Loewenstein D. Depression and risk for Alzheimer disease: systematic review, meta-analysis, and metaregression analysis. Arch Gen Psychiatry. 2006 May;63(5):530-8. doi: 10.1001/archpsyc.63.5.530. PMID 16651510
- [Background] Palmer K, Di Iulio F, Varsi AE, Gianni W, Sancesario G, Caltagirone C, Spalletta G. Neuropsychiatric predictors of progression from amnestic-mild cognitive impairment to Alzheimer's disease: the role of depression and apathy. J Alzheimers Dis. 2010;20(1):175-83. doi: 10.3233/JAD-2010-1352. PMID 20164594
- [Background] Pelton GH, Harper OL, Tabert MH, Sackeim HA, Scarmeas N, Roose SP, Devanand DP. Randomized double-blind placebo-controlled donepezil augmentation in antidepressant-treated elderly patients with depression and cognitive impairment: a pilot study. Int J Geriatr Psychiatry. 2008 Jul;23(7):670-6. doi: 10.1002/gps.1958. PMID 18088076
- [Background] Peskind ER, Potkin SG, Pomara N, Ott BR, Graham SM, Olin JT, McDonald S. Memantine treatment in mild to moderate Alzheimer disease: a 24-week randomized, controlled trial. Am J Geriatr Psychiatry. 2006 Aug;14(8):704-15. doi: 10.1097/01.JGP.0000224350.82719.83. PMID 16861375
- [Background] Petersen RC, Smith GE, Waring SC, Ivnik RJ, Tangalos EG, Kokmen E. Mild cognitive impairment: clinical characterization and outcome. Arch Neurol. 1999 Mar;56(3):303-8. doi: 10.1001/archneur.56.3.303. PMID 10190820
- [Background] Petersen RC, Thomas RG, Grundman M, Bennett D, Doody R, Ferris S, Galasko D, Jin S, Kaye J, Levey A, Pfeiffer E, Sano M, van Dyck CH, Thal LJ; Alzheimer's Disease Cooperative Study Group. Vitamin E and donepezil for the treatment of mild cognitive impairment. N Engl J Med. 2005 Jun 9;352(23):2379-88. doi: 10.1056/NEJMoa050151. Epub 2005 Apr 13. PMID 15829527
- [Background] Porsteinsson AP, Grossberg GT, Mintzer J, Olin JT; Memantine MEM-MD-12 Study Group. Memantine treatment in patients with mild to moderate Alzheimer's disease already receiving a cholinesterase inhibitor: a randomized, double-blind, placebo-controlled trial. Curr Alzheimer Res. 2008 Feb;5(1):83-9. doi: 10.2174/156720508783884576. PMID 18288936
- [Background] Ramakers IH, Visser PJ, Aalten P, Kester A, Jolles J, Verhey FR. Affective symptoms as predictors of Alzheimer's disease in subjects with mild cognitive impairment: a 10-year follow-up study. Psychol Med. 2010 Jul;40(7):1193-201. doi: 10.1017/S0033291709991577. Epub 2009 Nov 11. PMID 19903364
- [Background] Reisberg B, Doody R, Stoffler A, Schmitt F, Ferris S, Mobius HJ; Memantine Study Group. Memantine in moderate-to-severe Alzheimer's disease. N Engl J Med. 2003 Apr 3;348(14):1333-41. doi: 10.1056/NEJMoa013128. PMID 12672860
- [Background] Reynolds CF 3rd, Butters MA, Lopez O, Pollock BG, Dew MA, Mulsant BH, Lenze EJ, Holm M, Rogers JC, Mazumdar S, Houck PR, Begley A, Anderson S, Karp JF, Miller MD, Whyte EM, Stack J, Gildengers A, Szanto K, Bensasi S, Kaufer DI, Kamboh MI, DeKosky ST. Maintenance treatment of depression in old age: a randomized, double-blind, placebo-controlled evaluation of the efficacy and safety of donepezil combined with antidepressant pharmacotherapy. Arch Gen Psychiatry. 2011 Jan;68(1):51-60. doi: 10.1001/archgenpsychiatry.2010.184. PMID 21199965
- [Background] Ritchie K, Artero S, Touchon J. Classification criteria for mild cognitive impairment: a population-based validation study. Neurology. 2001 Jan 9;56(1):37-42. doi: 10.1212/wnl.56.1.37. PMID 11148233
- [Background] Sachs-Ericsson N, Corsentino E, Moxley J, Hames JL, Rushing NC, Sawyer K, Joiner T, Selby EA, Zarit S, Gotlib IH, Steffens DC. A longitudinal study of differences in late- and early-onset geriatric depression: depressive symptoms and psychosocial, cognitive, and neurological functioning. Aging Ment Health. 2013;17(1):1-11. doi: 10.1080/13607863.2012.717253. Epub 2012 Aug 30. PMID 22934752
- [Background] Salloway S, Ferris S, Kluger A, Goldman R, Griesing T, Kumar D, Richardson S; Donepezil 401 Study Group. Efficacy of donepezil in mild cognitive impairment: a randomized placebo-controlled trial. Neurology. 2004 Aug 24;63(4):651-7. doi: 10.1212/01.wnl.0000134664.80320.92. PMID 15326237
- [Background] Steffens DC, Potter GG. Geriatric depression and cognitive impairment. Psychol Med. 2008 Feb;38(2):163-75. doi: 10.1017/S003329170700102X. Epub 2007 Jun 22. PMID 17588275
- [Background] Wilson RS, Barnes LL, Mendes de Leon CF, Aggarwal NT, Schneider JS, Bach J, Pilat J, Beckett LA, Arnold SE, Evans DA, Bennett DA. Depressive symptoms, cognitive decline, and risk of AD in older persons. Neurology. 2002 Aug 13;59(3):364-70. doi: 10.1212/wnl.59.3.364. PMID 12177369
- [Background] Winblad B, Gauthier S, Scinto L, Feldman H, Wilcock GK, Truyen L, Mayorga AJ, Wang D, Brashear HR, Nye JS; GAL-INT-11/18 Study Group. Safety and efficacy of galantamine in subjects with mild cognitive impairment. Neurology. 2008 May 27;70(22):2024-35. doi: 10.1212/01.wnl.0000303815.69777.26. Epub 2008 Mar 5. PMID 18322263
- [Background] Zarate CA Jr, Singh JB, Quiroz JA, De Jesus G, Denicoff KK, Luckenbaugh DA, Manji HK, Charney DS. A double-blind, placebo-controlled study of memantine in the treatment of major depression. Am J Psychiatry. 2006 Jan;163(1):153-5. doi: 10.1176/appi.ajp.163.1.153. PMID 16390905
- [Derived] Pelton GH, Harper OL, Roose SP, Marder K, D'Antonio K, Devanand DP. Combined treatment with memantine/es-citalopram for older depressed patients with cognitive impairment: a pilot study. Int J Geriatr Psychiatry. 2016 Jun;31(6):648-55. doi: 10.1002/gps.4375. Epub 2015 Nov 11. PMID 26559790

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 35 depressed and cognitively impaired patients were recruited from the Late Life Depression and Memory Disorders Clinic at Columbia University Medical Center.
Pre-assignment Details: Any patients who were diagnosed with schizophrenia, psychoses, bipolar disorder, or alcohol/substance dependence (within the last 6 months) were excluded from participating in the study. Patients already on an effective anti-depressant, non-responders to citalopram/es-citalopram, and those on cholinesterase inhibitors/memantine were also excluded.
Groups:
- Es-citalopram and Memantine Treatment: This group received concurrent es-citalopram plus memantine treatment for 48 weeks. Patients ranged in age from 50-90 years old. Es-citalopram treatment began at 10mg per day for two weeks and was increased to 20mg per day for the 48 week duration. If a patient had an inadequate response to the antidepressant on two consecutive visits, the study physician used an alternative. At two weeks into the study, the patients were started on memantine 5mg, and the maximum dose of 20mg was reached by the six week point.
Period: Overall Study
Arm/Group | Es-citalopram and Memantine Treatment
Started | 35
Completed | 26
Not Completed | 9
Not completed — Withdrawal by Subject | 5
Not completed — Physician Decision | 2
Not completed — Patients moved | 2

BASELINE CHARACTERISTICS:
Arm/Group | Es-citalopram and Memantine Treatment
Number analyzed (Participants) | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.3 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 28
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 35

OUTCOME MEASURES:

1. Primary Outcome: Change in Selective Reminding Test - Total Immediate Recall (SRT-IR)
Description: Change in Selective Reminding Test-Total Immediate Recall (SRT-IR) scores from baseline to Week 48: Measures word recall (maximum 12 words per trial, across 6 trials). Maximum total recall score across 6 trials is 72; minimum recall is 0 across 6 trials. The higher the raw score, the better the patient did at recalling the target words. The unit of measure is the raw score, or the sum of the number of words recalled across all 6 trials.
Time Frame: baseline, 48 weeks
Population: Analysis was intent to treat.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Es-citalopram and Memantine Treatment
Number analyzed (Participants) | 35
units on a scale | 7.5 (15)

2. Secondary Outcome: Change in Wechsler Memory Scale-III (WMS-III)
Description: Change in Wechsler Memory Scale-III scores from baseline to Week 48: The WMS-III Visual Reproduction sub-test was used to measure visual working memory and delayed memory. Patients were shown pictures of four drawings and were asked to reproduce them from memory immediately after seeing them, and 25 minutes after seeing them. The four scores are summed and the greater the total raw score, the better the patient did on the assessment. The maximum raw score for this test is a 41 on both the immediate and delayed portions (the overall range is 0-82 points). The change score is calculated using the total scores of both the immediate and delayed portions.
Time Frame: Baseline, Week 48
Population: Analysis was intent to treat.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Es-citalopram and Memantine Treatment
Number analyzed (Participants) | 35
units on a scale | 9.9 (32.8)

3. Secondary Outcome: Change in Selective Reminding Test - Delayed Recall (SRT-DR)
Description: Change in Selective Reminding Test-Delayed Recall scores from baseline to Week 48: SRT Delay is administered 15 minutes after the immediate recall portion. Patients are asked to remember as many of the words as they can from the 6 trials. Maximum raw score is a 12 for free recall. If a patient is unable to recall a word, they are given a chance to recognize it among three incorrect word choices. Maximum raw score for recognition is 12. The greater the score on the delayed recall portion, the better the patient does on the assessment.
Time Frame: Baseline, Week 48
Population: Analysis was intent to treat.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Es-citalopram and Memantine Treatment
Number analyzed (Participants) | 35
units on a scale | 1.2 (3.9)

4. Secondary Outcome: Change in Trails B
Description: Change from baseline to Week 48 on Trails B: Measures attention and executive function. It asks patients to connect numbers and letters in numerical to alphabetical order from (1-13 and A-L) as fast as they can. Patients are timed; the longer it takes for the patient to connect the numbers and letters, the worse their score. Unit of measure is in seconds. The amount of errors that the patient makes during trails is also recorded.
Time Frame: Baseline, Week 48
Population: Analysis was intent to treat.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Es-citalopram and Memantine Treatment
Number analyzed (Participants) | 35
seconds | -36.3 (74.5)

5. Secondary Outcome: Change in Trails A
Description: Change in Trails A scores from baseline to Week 48: Measures attention and executive function. It asks patients to connect numbers from 1-25 in numerical order as fast as they can. Patients are timed; the longer it takes for the patient to connect the numbers, the worse their score. Unit of measure is in seconds. The amount of errors that the patient makes during trails is also recorded.
Time Frame: Baseline, Week 48
Population: Analysis was intent to treat.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Es-citalopram and Memantine Treatment
Number analyzed (Participants) | 35
seconds | 1.9 (41.2)

6. Other Pre Specified Outcome: Change in 24-item HAMD
Description: Change in 24-item Hamilton Rating Scale for Depression (HAMD) scores from baseline to Week 48: HAMD measures depression severity based on a series of 24 items items. The range of HAMD total score is 0-74; 0 indicates no depressive symptoms and a maximum HAMD score is a 74, where the greater the score indicates more significant psychopathology. In this study, moderate to severe depression is considered a HAMD-24 greater than 14.
Time Frame: Baseline, Week 48
Population: Analysis was intent to treat.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Es-citalopram and Memantine Treatment
Number analyzed (Participants) | 35
scores on a scale | -15.2 (4.4)

7. Other Pre Specified Outcome: Change in Treatment Emergent Side Effects (TESS)
Description: Somatic side effect rating scale which includes 26 common somatic side effects associated with previous medication clinical trials; rated by the study physician. Factors were dichotomized to "yes" or "no" responses on this scale, which equated to the symptom being either present or not present. "Yes" and "no" responses were given a value of 0 (no) or 1 (yes). Responses from the entire group were calculated and the mean at baseline and the last visit is reported below.
Time Frame: Baseline, Week 48
Population: Analysis was intent to treat.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Es-citalopram and Memantine Treatment
Number analyzed (Participants) | 35
units on a scale
  Treatment Emergent Side Effects (Baseline) | 6.6 (4.2)
  Treatment Emergent Side Effects (WK 48) | 3.2 (2.9)

8. Other Pre Specified Outcome: Change in Clinical Global Impression - Depression Change
Description: The CGI Depression Change follows a seven-point likert scale. Compared to the patient's condition at baseline in the study [prior to medication initiation], the patient's condition is rated as: 1=very much improved since the initiation of treatment; 2=much improved; 3=minimally improved; 4=no change from baseline (the initiation of treatment); 5=minimally worse; 6= much worse; 7=very much worse since the initiation of treatment. Responses were calculated for the entire group. Mean at final visit has been reported below. Higher mean at baseline indicates a decrease in depression scores.
Time Frame: Baseline, Week 48
Population: Analysis was intent to treat; ANOVA repeated measures. All values of data collected were included, except for those who exited the study early. In these cases, their last observation was carried forward (LOC).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Es-citalopram and Memantine Treatment
Number analyzed (Participants) | 35
units on a scale
  Cognitive Global Impression at Baseline | 4.1 (0.5)
  Cognitive Global Impression at Final Visit (WK 48) | 2.1 (1.2)

9. Other Pre Specified Outcome: Change in Clinical Global Impression - Cognitive Change
Description: The CGI Cognitive Change follows a seven-point likert scale. Compared to the patient's condition at baseline in the study [prior to medication initiation], the patient's condition is rated as: 1=very much improved since the initiation of treatment; 2=much improved; 3=minimally improved; 4=no change from baseline (the initiation of treatment); 5=minimally worse; 6= much worse; 7=very much worse since the initiation of treatment. Responses from the entire group were calculated. Mean at final visit and baseline is reported below.
Time Frame: Baseline, Week 48
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Es-citalopram and Memantine Treatment
Number analyzed (Participants) | 35
units on a scale
  CGI-Cognitive Change (Baseline) | 3.6 (0.6)
  Clinical Global Impression-Cogntive Change (WK 48) | 2.7 (0.9)

10. Other Pre Specified Outcome: Conversion to Dementia Using Clinical Dementia Rating (CDR)
Description: The CDR is a numeric rating scale that is used to quantify the severity of one's cognitive function. The scale goes from 0=normal; 0.5=mild cognitive impairment; 1 to 3=mild to moderate/severe dementia. CDR was used a dichotomous outcome measure (no=0; yes=1).
Time Frame: Baseline, Week 48
Population: as for outcome 8
Measure: Number; unit: participants
Arm/Group | Es-citalopram and Memantine Treatment
Number analyzed (Participants) | 35
participants | 1

ADVERSE EVENTS:
Time Frame: From initiation of study until one month after study completion- a total of 13 months.
Arm/Group | Es-citalopram and Memantine Treatment
Serious Adverse Events (participants affected / at risk) | 2/35
Other Adverse Events (participants affected / at risk) | 4/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Es-citalopram and Memantine Treatment (N=35)
Syncopal Episode (Cardiac disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Es-citalopram and Memantine Treatment (N=35)
Headache (Nervous system disorders) | 1 (4)
Sedation (Nervous system disorders) | 2 (4)
Nausea (Gastrointestinal disorders) | 1 (4)

LIMITATIONS AND CAVEATS:
* The inclusion criteria required all patients to have an MMSE of 24 or higher, which may have lowered the conversion rate to dementia
* small sample size
* cognitive improvement may have been due in part to combined es-citalopram and memantine

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No